CLINICAL TRIAL: NCT05931432
Title: A Tailored and Digital Approach to Address Equity and Support Well-being for Healthcare Workers in the Era of COVID
Acronym: Thrive
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 852022
Record Dates: First submitted 2023-05-16; First posted 2023-07-05 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Depression, Anxiety; Satisfaction; Well-being
MeSH Terms: conditions — Depression; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants will be asked to complete an ICF and baseline survey at enrollment. They will be given survey assessments at 0, 18 and 30 months. Survey assessments will include validated measures on well-being, depression, anxiety, stress, resilience, and job satisfaction of physicians.
  The control group will have access to usual care well-being resources at Penn Medicine. These include links, classes, groups, social media sites such as Penn Cobalt which require self-awareness to find the resources and access them. In this context, the individual has to "pull" the resources they need and there may be several barriers to completing each step
- Comprehensive Well-Being Intervention (Experimental): Participants will be asked to complete an ICF and baseline survey at enrollment. Participants will complete a full assessment using validated instruments at enrollment, 18 months and 30 months (depression, anxiety, stress, resilience, and job satisfaction). Participants will also complete the brief well-being index (WBI, nine questions) every 3 months over 30 months. The primary endpoint is assessed at 18 months. A secondary endpoint of persistence of effect is measured at 30 months.
  The intervention group will receive an 18-month comprehensive suite of services including: 1) monthly automated text messaging reminders about wellbeing resources focused on a range of topics (e.g. mindfulness, stress management, childcare support, racial trauma, diversity and inclusion) and assignment to a one-hour quarterly peer support group with an expectation of regular attendance. Half of these sessions will be self-directed discussion topics and half will be facilitated discussions.
  Interventions: Other: Comprehensive Well-Being Intervention

INTERVENTIONS:
Other: Comprehensive Well-Being Intervention — The intervention group will receive an 18-month comprehensive suite of services including: 1) monthly automated text messaging reminders about wellbeing resources focused on a range of topics (e.g. mindfulness, stress management, childcare support, racial trauma, diversity and inclusion) and assignment to a one-hour quarterly peer support group with an expectation of regular attendance. Half of these sessions will be self-directed discussion topics and half will be facilitated discussions. The content of monthly text messaging resources and discussion topics for the peer-support groups will be informed by the Aim 1 qualitative findings.
  Arms: Comprehensive Well-Being Intervention

SUMMARY:
For this project the broad research objective is to evaluate the effectiveness of an enhanced digital wellbeing program in improving well-being, depression, anxiety, stress, resilience, and job satisfaction of physicians. The intent of the investigators is that this will enable a proactive culture of well-being and mental health support for the broader healthcare workforce during the multiple phases of the pandemic.

The investigator's approach evaluates existing digital models which can be executed in a timely fashion and rapidly scaled for use across other health systems.

Aim 1: Conduct interviews of URM and women physicians to identify barriers and facilitators to accessing and receiving digital well-being, mental health, and culturally sensitive support resources.

Aim 2: Through a randomized controlled trial (RCT) investigate the immediate and long-term effect of a comprehensive well-being focused intervention (push text messaging, resource support, semi-facilitated peer groups hosted by Cobalt) vs. usual care on well-being, depression, anxiety, stress, resilience, and job satisfaction of physicians practicing in the era of COVID.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age;
* Interest in participating in an 18 month study and willing to complete regular surveys;
* Regular, daily access to a phone with texting capabilities
* Identify as a Physician at Penn Medicine;

Exclusion Criteria:

* Under 18 years of age;
* Not willing to sign informed consent document for an 18 month study;
* No access to a phone with texting capabilities;
* Not a Physician at Penn Medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-07-27 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Well-Being Index (WBI) | at month 0
  The Well-being index (WBI) is a nine-question survey validated for use in physician populations and considered important to health systems in managing the well-being of their workforce. The domains address likelihood of burnout, severe fatigue, suicidal ideation, quality of life, meaning in work, work-life integration, risk of medical error, dropout risk, and overall well-being, It is brief (approximately 5 minutes to complete), easily tracked via a mobile app, and tracked across multiple health systems in Pennsylvania and across the United States. The WBI is also currently used by our health system for assessing HCW well-being and baseline survey
Well-Being Index (WBI) | at month 3
  The Well-being index (WBI) is a nine-question survey validated for use in physician populations and considered important to health systems in managing the well-being of their workforce. The domains address likelihood of burnout, severe fatigue, suicidal ideation, quality of life, meaning in work, work-life integration, risk of medical error, dropout risk, and overall well-being, It is brief (approximately 5 minutes to complete), easily tracked via a mobile app, and tracked across multiple health systems in Pennsylvania and across the United States. The WBI is also currently used by our health system for assessing HCW well-being and baseline survey
Well-Being Index (WBI) | at month 6
  The Well-being index (WBI) is a nine-question survey validated for use in physician populations and considered important to health systems in managing the well-being of their workforce. The domains address likelihood of burnout, severe fatigue, suicidal ideation, quality of life, meaning in work, work-life integration, risk of medical error, dropout risk, and overall well-being, It is brief (approximately 5 minutes to complete), easily tracked via a mobile app, and tracked across multiple health systems in Pennsylvania and across the United States. The WBI is also currently used by our health system for assessing HCW well-being and baseline survey
Well-Being Index (WBI) | at month 9
  The Well-being index (WBI) is a nine-question survey validated for use in physician populations and considered important to health systems in managing the well-being of their workforce. The domains address likelihood of burnout, severe fatigue, suicidal ideation, quality of life, meaning in work, work-life integration, risk of medical error, dropout risk, and overall well-being, It is brief (approximately 5 minutes to complete), easily tracked via a mobile app, and tracked across multiple health systems in Pennsylvania and across the United States. The WBI is also currently used by our health system for assessing HCW well-being and baseline survey
Well-Being Index (WBI) | at month 12
  The Well-being index (WBI) is a nine-question survey validated for use in physician populations and considered important to health systems in managing the well-being of their workforce. The domains address likelihood of burnout, severe fatigue, suicidal ideation, quality of life, meaning in work, work-life integration, risk of medical error, dropout risk, and overall well-being, It is brief (approximately 5 minutes to complete), easily tracked via a mobile app, and tracked across multiple health systems in Pennsylvania and across the United States. The WBI is also currently used by our health system for assessing HCW well-being and baseline survey
Well-Being Index (WBI) | at month 15
  The Well-being index (WBI) is a nine-question survey validated for use in physician populations and considered important to health systems in managing the well-being of their workforce. The domains address likelihood of burnout, severe fatigue, suicidal ideation, quality of life, meaning in work, work-life integration, risk of medical error, dropout risk, and overall well-being, It is brief (approximately 5 minutes to complete), easily tracked via a mobile app, and tracked across multiple health systems in Pennsylvania and across the United States. The WBI is also currently used by our health system for assessing HCW well-being and baseline survey

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-2) | at month 0
  PHQ-2 and GAD-2 have been validated and used in multiple studies and provide easy, simple scales to quickly assess for depression and anxiety.
Patient Health Questionnaire (PHQ-2) | at month 18
  PHQ-2 and GAD-2 have been validated and used in multiple studies and provide easy, simple scales to quickly assess for depression and anxiety.
General Anxiety Disorder (GAD-2) | at month 0
  GAD-2 have been validated and used in multiple studies and provide easy, simple scales to quickly assess for depression and anxiety. GAD-2 have been validated and used in multiple studies and provide easy, simple scales to quickly assess for depression and anxiety.
General Anxiety Disorder (GAD-2) | at month 18
  GAD-2 have been validated and used in multiple studies and provide easy, simple scales to quickly assess for depression and anxiety. GAD-2 have been validated and used in multiple studies and provide easy, simple scales to quickly assess for depression and anxiety.
Perceived Stress Scale (PSS-10) | at month 0
  The Perceived Stress Scale is a 10-item well validated instrument in physician cohorts and measures stress
Perceived Stress Scale (PSS-10) | at month 18
  The Perceived Stress Scale is a 10-item well validated instrument in physician cohorts and measures stress
Connor-Davidson Resilience Scale (CDRS) | at month 0
  The Connor-Davidson Resilience Scale (CDRS) is a 2-item standardized and validated instrument in physician populations and measures bounce back and adaptability aspects of resilience
Connor-Davidson Resilience Scale (CDRS) | at month 18
  The Connor-Davidson Resilience Scale (CDRS) is a 2-item standardized and validated instrument in physician populations and measures bounce back and adaptability aspects of resilience
Physician Job Satisfaction Scale (JSS-10) | at month 0
  The Physician Job Satisfaction Scale (JSS-10) measures satisfaction at work and is a well validated 12-item measure
Physician Job Satisfaction Scale (JSS-10) | at month 18
  The Physician Job Satisfaction Scale (JSS-10) measures satisfaction at work and is a well validated 12-item measure
Professional Fulfillment Index | at month 0
  • The Professional Fulfillment Index (PFI) was developed to capture both burnout and professional fulfillment in the evaluation and assessment of professional wellbeing [18]. The PFI is a 16-item index that measures burnout and professional fulfillment.
Professional Fulfillment Index | at month 18
  • The Professional Fulfillment Index (PFI) was developed to capture both burnout and professional fulfillment in the evaluation and assessment of professional wellbeing [18]. The PFI is a 16-item index that measures burnout and professional fulfillment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States